# Feasibility Study of a Behavioral Parent Intervention to Support Selfmanagement in Pediatric Typ 1 Diabetes: Statistical Analysis Plan

Version 1, date 2025-01-10

### ClinicalTrials.gov registration:

First published in ClinicalTrials.gov 09/16/2024 (ID: NCT06599840).

#### **Ethics consent:**

Approved by the Swedish Ethical Review Authority 24/05/2021 (No 2021-01558). Amendments approved 10/07/2024 (No 2024-04149-02) and 29/09/2024 (No 2024-05953-02).

# **Principal Investigator:**

Brjánn Ljótsson, PhD, professor Department of Clinical Neuroscience, Division of Psychology Nobels väg 9, 17176 Karolinska Institute, Stockholm, Sweden E-mail: brjann.ljotsson@ki.se, Telephone: +46 (0)739823884

# Feasibility criteria

- 1) Participation: at least 70% of participants or their partners attend at least four of the six initial sessions.
- 2) Satisfaction: participants are satisfied with the program's structure and content by scoring a mean of at least 24 points on the Client Satisfaction Questionnaire.
- 3) Engagement in the six behavioral assignments that are presented at each of the first six weeks' sessions as "this week's tool". Engagement is measured by weekly parent reports of 1) **frequency:** how often they used it (0-7 points reflecting number of days used), 2) **intensity**: how much effort they have put down in using it (0 = none, to 5 = a lot) and 3) **usability:** how helpful they perceive the strategy to be for them (0 = not at all, to 5 = very). We have chosen feasibility criteria to be met if mean scores for the whole group and all the components exceed 2 points in each of the three domains. The score will also be calculated separately for each component to investigate need of adjustments or removal of specific modules.
- 4) Whether the set of questionnaires is of reasonable size and capture relevant parameters according to the participants. Perception of questionnaire size is measured by asking participating parents to score how much time they perceived the questionnaires took ranging from 1-4 points (1 = a short while, 2 = reasonably long time, 3 = long time but it felt OK, 4 = too much time) after finishing the T2 questionnaires. This is followed by the same question regarding the weekly questionnaires. Children will answer the same question at the end of the T2 questionnaires. A mean score will be calculated for each of the assessments (T2 for parents, T2 for children, and weekly measurements for parents) and a score below 3 will be considered as reasonable questionnaire size. Perception of relevance is measured by asking participating parents whether the questions have captured relevant aspects rated from 1-4 (1 = yes totally, 2 = to a large extent, 3 = to some extent, 4 = not at all). This question is not posed to the children as it is considered difficult for a child to answer. If the mean score is 2,5 or less the questionnaires is considered to capture relevant aspects according to the participants.

### Assessments

Outcome measures are assessed at three main time points: T1) baseline: one week before the intervention starts, T2) primary end point: four weeks after the last session, and T3) at 3-month follow-up: three months after primary end point. To explore change over the course of the intervention and mediators of change, a subset of the outcome variables are assessed weekly or every second week during the 15 weeks between baseline and primary endpoint. See table 1 for a full list of variables.

# Statistical analysis of potential effects

Analysis of outcomes are performed using linear mixed models with time as independent variable, coded as a factor with two levels (T2 and T3) and baseline (T1) as the reference value. Secondary moderation analyses will be conducted to explore if ADHD symptoms in children and participating parents predict change on the primary outcome variable. The moderation analysis will be performed on the weekly collected outcome during treatment to optimize statistical power.

Within-group mediation analysis will be conducted using linear mixed models to investigate whether changes over time in diabetes treatment satisfaction, TiT and the parent-reported percentage of times their children have taken insulin and reacted to low / high blood glucose levels out of all the times it has been needed during the last week ("Getting Self-Management Routines Done") are mediated by a change in parent-reported behavioral challenges in diabetes self-management, as measured by a non-validated questionnaire newly developed by the research group (Parental Challenges in Diabetes Self-Management).

# Thematic analysis of interview data

Shortly after the sixth session, parents will be asked to participate in a short telephone interview conducted by psychology students with T1D knowledge, answering open-ended questions on their experiences of the intervention. Qualitative analysis of interview data will be performed with reflexive thematic analysis.

Table 1. Variables, measurements, and their assessment time points.

| | Variable | Measurement | Assessment time points |
|---|---|---|---|
| Parent-<br>reported<br>data | Diabetes treatment satisfaction (primary outcome measure) | Diabetes Treatment Satisfaction Questionnaire (DTSQ) | T1,T2, T3,<br>weekly<br>assessments<br>between T1-T2 |
| | Self-management behaviors (proxy) | Getting Self-Management Routines Done | |
| | Parental challenges in diabetes self-<br>management | Parental Challenges in Diabetes Self-Management | |
| | Parents' symptoms of anxiety | General Anxiety Disorder – 7 (GAD-7) | |
| | Child ADHD symptoms | ADHD Self Report Scale for Parents (ASRS) | T1 |
| | Parent ADHD symptoms | Adult ADHD Self-Report Scale (A-ASRS) | |
| | Satisfaction with intervention | Client Satisfaction Questionnaire (CSQ) | T2 |
| | Diabetes related family conflicts | Diabetes Family Conflict Scale (DFCS) – parent report | T1, T2, T3 |
| | Parents' symptoms of stress | Perceived Stress Scale (PSS) | |
| | Parenting behaviors | Parenting Practices Scale | |
| | Parent self-efficacy | Me As Parent | |
| | Parent quality of life | Peds Quality of Life - Family Impact Measure (PedsQL-FIM) | |
| | Child health related quality of life | DISABKIDS – generic module, parent report | |
| Child-<br>reported<br>data | Child health related quality of life | DISABKIDS – generic module and diabetes module, child report | T1, T2 |
| | Diabetes related family conflicts | Diabetes Family Conflict Scale (DFCS), youth report | |
| Medical data<br>from NDR | Glycemic control | Glycated haemoglobin (HbA1c) | Closest before T1, after T2 and T3 |
| | Physical activity | Number of days a week being physically active | Closest before T1, after T3 |
| | Appointments at the diabetes clinic | Number of diabetes clinic appointments | |
| | Ketoacidosis | Incidents of ketoacidosis | |
| | Severe hypoglycaemia | Incidents of severe hypoglyceamia | |
| Medical data<br>from online<br>glucose<br>system<br>Glooko | Time in target | % time blood glucose values are within the target interval 4-8 mmol/mol the last 2 weeks | T1, T2, T3,<br>assessments<br>every second<br>week between<br>T1-T2 |
| | Time with low blood glucose | % time blood glucose values are below 3 mmol/mol the last 2 weeks | |
| | Time with high blood glucose | % time blood glucose values are above 12,9 mmol/mol the last 2 weeks | |
| | Mean blood glucose | Mean blood glucose value the last 2 weeks | |
| | Blood glucose variation | Standard deviation of blood glucose values the last 2 weeks | |

T1: baseline assessment, T2: primary end point assessment, T3: three months follow-up assessment.